CLINICAL TRIAL: NCT07120022
Title: Training Cold Showers: A Randomized Controlled Study
Brief Title: Self-efficacy Training to Facilitate Taking Cold Showers
Acronym: TCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: eknz2023-01677
Record Dates: First submitted 2025-07-22; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Psychological and Behavioral Symptoms
MeSH Terms: conditions — Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-efficacy training (Experimental): Self-efficacy training
  Interventions: Other: Self-efficacy training
- No Training (No Intervention): No Training

INTERVENTIONS:
Other: Self-efficacy training — The primary goal of this study is to determine whether self-efficacy training can increase the probability of taking cold showers regularly over a three-month period.
  Arms: Self-efficacy training

SUMMARY:
The primary goal of this study is to determine whether a self-efficacy training can increase the probability of taking cold showers regularly over a three-month period. Secondary objectives are to assess effects on physical and mental well-being, sleep quality, skin and hair appearance, perceived illness, and related sickness absences from work.

DETAILED DESCRIPTION:
This study is an extension of our two ongoing studies: Feasibility and effects of taking cold showers: A randomized controlled study (Study ID 2019-00529) and Mindset interventions to facilitate taking cold showers: A randomized controlled study (Study ID 2022-00952), which have been approved by the EKNZ. Our ongoing study closely follows the protocol of a previous and similar study by Buijze and colleagues (2016).

This study extends our ongoing study by including experimental conditions, while retaining the original study procedure, i.e., the same recruitment, inclusion/exclusion criteria, and assessments.

ELIGIBILITY:
Inclusion criteria

* In good health and between 18 and 65 years of age
* Do not take cold showers on a regular basis

Exclusion criteria

* Pregnant or lactating women (assessed via self-report)
* Cardiac, pulmonary or any other severe disease (assessed via self-report)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Showering behaviour concerning frequency (Baseline) | Baseline
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Baseline) | Baseline
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Baseline) | Baseline
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 1) | Week 1
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 1) | Week 1
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 1) | Week 1
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 2) | Week 2
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 2) | Week 2
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 2) | Week 2
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 3) | Week 3
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 3) | Week 3
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 3) | Week 3
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 4) | Week 4
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 4) | Week 4
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 4) | Week 4
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 5) | Week 5
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 5) | Week 5
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 5) | Week 5
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 6) | Week 6
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 6) | Week 6
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 6) | Week 6
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 7) | Week 7
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 7) | Week 7
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 7) | Week 7
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 8) | Week 8
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 8) | Week 8
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 8) | Week 8
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 9) | Week 9
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 9) | Week 9
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 9) | Week 9
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 10) | Week 10
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 10) | Week 10
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 10) | Week 10
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 11) | Week 11
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 11) | Week 11
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 11) | Week 11
  Participants will be asked their motivation for taking cold showers during the last week.
Showering behaviour concerning frequency (Week 12) | Week 12
  Participants will be asked how often they showered during the last week.
Showering behaviour concerning duration (Week 12) | Week 12
  Participants will be asked how long they showered for during the last week.
Showering behaviour concerning motivation (Week 12) | Week 12
  Participants will be asked their motivation for taking cold showers during the last week.

SECONDARY OUTCOMES:
WHO Five Well-Being Index | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The WHO-5 is a short questionnaire designed to measure well-being. The WHO-5 consists of five questions. The answers are given on a six-level scale (0 - 5, where 0 represents "No time at all" and 5 "All the time"). The raw value is obtained by adding the answers. The raw value ranges from 0 to 25, where 0 is the lowest quality of life and 25 is the highest quality of life. The percentage value of 0 -100 is obtained by multiplying by 4. The percentage value 0 denotes the worst state of health, 100 the best. The processing time is less than one minute. Example: In the last 4 weeks I was happy and in a good mood.
Questionnaire for positive aspects of well-being in adults | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The FEW 16 is a psychological self-evaluation procedure for the assessment of positive aspects of well-being in adults. The FEW 16 consists of 16 questions, of which 4 questions each are assigned to one of the following four scales: Ability to work under pressure, vitality, enjoyment, inner peace. The answers are given on a 6-level scale (1 - 6, where 6 represents "Does not apply at all" and 1 "Is absolutely true"). The processing time is estimated at five to ten minutes by adding up the 16 items you get an overall result between 16 - 96, whereas a lower overall result shows a higher physical wellbeing. Example: There's hardly anything that can upset me.
International Physical Activity Questionnaire | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The IPAQ is a short questionnaire designed to measure physical activity. The IPAQ consists of six questions, of which 3 questions each are assigned to one of the following two scales: Strong physical exertion and light physical exertion. Either you have to tick an answer or you will be asked for a time in hours and minutes per week. The processing time is estimated at three minutes. Example: If you are thinking about physical activities where you are at least a little out of breath, such as running, hiking, dancing, gardening or many sports, how many days a week do you do physical activities of this kind?
Pittsburgh Sleep Quality Index | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. The questionnaire offers seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totalling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Example: How tired are you during the day?
Skin quality questionnaire | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  The SQQ is a short self-report questionnaire that assesses hand and skin quality. The measure consists of 4 items, whereas they measure appearance, intactness, moisture content and sensation on a 7-level scale (1-7), where higher scores denote a healthier quality of skin. The processing time is less than one minute each. Example: Appearance: Abnormal: redness, stains, rash. Normal: no redness, stains or rashes.
Sickness absence and illness days | All secondary outcomes will be assessed at baseline and then monthly for 3 months.
  Will be assessed at baseline and then monthly for 3 months. Participants are asked to retrospectively indicate the total number of days of absence from their work due to sickness and to indicate the number of days that they have had symptoms of illness, cold or flu during the last month. If participants indicate sickness absence or illness over five days, they are asked for the reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof. Dr., Principal Investigator — University of Basel, Division Clinical Psychology and Psychotherapy
Locations (1):
- University of Basel Faculty of Psychology Division for Clinical Psychology and Psychotherapy, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buijze GA, Sierevelt IN, van der Heijden BC, Dijkgraaf MG, Frings-Dresen MH. The Effect of Cold Showering on Health and Work: A Randomized Controlled Trial. PLoS One. 2016 Sep 15;11(9):e0161749. doi: 10.1371/journal.pone.0161749. eCollection 2016. PMID 27631616